CLINICAL TRIAL: NCT05294484
Title: Study on the Effect of Genetic Polymorphisms of Uridine Diphosphate Glucuronosyl Transferase (UGT) on the Pharmacokinetics of Indapamide in Egyptians
Brief Title: Effect of Genetic Polymorphisms of UGT on the PKs of Indapamide in Egyptians
Acronym: UGT/PKs
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PG/PK Study on Indapamide
Record Dates: First submitted 2021-08-10; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2021-12

CONDITIONS: Pharmacogenomics
MeSH Terms: interventions — Indapamide

STUDY DESIGN:
Intervention Model Description: A comparative randomized, single-dose, two-treatment (fed vs. fasting), parallel design of indapamide in healthy adult Egyptions
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fasting group (Active Comparator): Following an overnight fast of at least 10 hours, subjects should be administered single dose of indapamide 1.5 mg SR with 240 mL (8 fluid ounces) of water. No food should be allowed for at least 4 hours post-dose. Water can be allowed as desired except for one hour before and after drug administration. Subjects should receive standardized meals scheduled at the same time in each period of the study.
  Interventions: Drug: Indapamide 1.5 MG SR
- Fed group (Active Comparator): Following an overnight fast of at least 10 hours, subjects should start the recommended meal 30 minutes prior to administration of the drug. Study subjects should eat this meal in 30 minutes or less; however, indapamide 1.5 mg SR should be administered 30 minutes after start of the meal. The drug should be administered with 240 mL (8 fluid ounces) of water. No food should be allowed for at least 4 hours post-dose. Water can be allowed as desired except for one hour before and after drug administration. Subjects should receive standardized meals scheduled at the same time in each period of the study.
  All subjects should abstain from the consumption of fruit juices during the study period. All the subjects are to be under complete medical supervision.
  Interventions: Drug: Indapamide 1.5 MG SR

INTERVENTIONS:
Drug: Indapamide 1.5 MG SR — the effect of genetic variation of UGT2B7 on human response to treatment with indapamide and its correlation with pharmacokinetic parameters in Egyptian subjects

SUMMARY:
The aim of this works is to investigate the effect of genetic variation of UGT2B7 on human response to treatment with indapamide and its correlation with pharmacokinetic parameters in Egyptian subjects.

DETAILED DESCRIPTION:
Indapamide is a thiazide-type diuretic commonly prescribed to treat mild to moderate hypertension. As it has fewer side effects in inducing metabolic derangements than other thiazide diuretics, indapamide is well accepted to be used as initial therapy to treat hypertension in patients with previous stroke or older people (over 80) or as an add-on treatment. However, severe hyponatremia and hypokalemia have been reported. Therefore, limiting the dose to that necessary to achieve maximal blood pressure reduction and improved cardiovascular outcomes is relevant. Although the major metabolites of indapamide have been identified, the pathways of cytochrome P450 (CYP450)-catalyzed indapamide biotransformation have not been fully elucidated. One recent report suggested that CYP2C19, CYP2C8, and CYP3A4 are involved in the metabolism. Recent advancement in the field of glucuronidation has identified a high degree of allelic diversity for human uridine diphosphate glucuronosyl transferases (UGTs).

As indapamide is glucuronidated by UGT enzymes, poly-morphisms in the genes encoding these drug-metabolizing enzymes could potentially influence its PK. Large inter-individual variability in the rate of glucuronidation of various drugs has been reported. The UGT2B7 enzyme is expressed in the liver and many extrahepatic tissues. Mutations in the UGT2B7 gene may therefore have pharmacological, toxicological, and physiological significance.

the investigators have little information on pharmacogenetics (PG) studies of indapamide. The effect of genetic variation on DMEs activity and the clinical impact on indapamide in particular are not fully understood.

The ultimate goal of personalized medicine is to identify specific genetic features with the differential risk of human diseases or the efficacy of certain therapeutic interventions . Mounting evidence has linked the genetic make-up to a significant portion of drug-induced toxicity. The primary focus of PG is DMEs activity.

The pharmacology of drugs subject to inherited variability in metabolism is often complex. Few have simple or single pathway of elimination. In addition, ethnicity may account for the observed differences in both pharmacokinetics (PK) and pharmacodynamics of drugs, thus resulting in variability in response to drug therapy. Furthermore, genetic polymorphism is one of the most important factors that may contribute to the ethnic sensitivity of a drug in its metabolic pathways.

Single nucleotide polymorphism (SNP) is the most frequently observed mutation in all organisms. The cost for mapping of the genetic variance among thousands of SNPs could be extremely high. Recent advances in whole-genome sequencing (WGS) have led to burst of bioinformation and a significant knowledge base for investigating the genetic architecture of drug metabolisms and treatment efficacies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should be healthy adult volunteers with age between (18-45) with normal body weight.
* The volunteers will be asked to provide a complete medical history, and complete a physical examination, laboratory tests (hematology, clinical chemistry, urinalysis, serology (including hepatitis B surface antigen, anti-hepatitis C virus and antihuman immunodeficiency virus antibody)

Exclusion Criteria:

* Treatment with any known enzyme -inducing /inhibiting agent within 30 days prior to the start of the study and throughout the study.
* Subjects who have taken any medication less than two weeks of the trials starting date
* Susceptibility to allergic reaction to study drugs
* Any prior surgery of the gastrointestinal tract that may interfere with drug absorption
* Gastrointestinal diseases
* Renal diseases
* Pancreatic disease including diabetes
* Hepatic diseases
* Hematological diseases or pulmonary diseases
* Abnormal laboratory values
* Subject who have donated blood or who have been involved in multiple dosing study requiring a large volume of blood (more than 500 ml) to be drawn within 6 weeks preceding the start of the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-03-15 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
the PK parameters of Indapamide following single oral dose include: | at Day 0: prior to drug administration (blank), then samples (5ml each) will be obtained at 0.5 hour, 1 hour, 1.5 hour, 2 hour, 2.5 hour, 3 hour, 4 hour, 5 hour, 6 hour, 8 hour, 10 hour, 12 hour, and 24 hour after drug administration
  area under the concentration-time curve over the dosing interval (AUC[0-tau])
maximum concentration (Cmax) | at Day 0: prior to drug administration (blank), then samples (5ml each) will be obtained at 0.5 hour, 1 hour, 1.5 hour, 2 hour, 2.5 hour, 3 hour, 4 hour, 5 hour, 6 hour, 8 hour, 10 hour, 12 hour, and 24 hour after drug administration
  maximum concentration (Cmax)
time of occurrence of Cmax (Tmax) | at Day 0: prior to drug administration (blank), then samples (5ml each) will be obtained at 0.5 hour, 1 hour, 1.5 hour, 2 hour, 2.5 hour, 3 hour, 4 hour, 5 hour, 6 hour, 8 hour, 10 hour, 12 hour, and 24 hour after drug administration
  time of occurrence of Cmax (Tmax)
terminal phase half-life (T1/2) | at Day 0: prior to drug administration (blank), then samples (5ml each) will be obtained at 0.5 hour, 1 hour, 1.5 hour, 2 hour, 2.5 hour, 3 hour, 4 hour, 5 hour, 6 hour, 8 hour, 10 hour, 12 hour, and 24 hour after drug administration
  terminal phase half-life (T1/2)
clearance | at Day 0: prior to drug administration (blank), then samples (5ml each) will be obtained at 0.5 hour, 1 hour, 1.5 hour, 2 hour, 2.5 hour, 3 hour, 4 hour, 5 hour, 6 hour, 8 hour, 10 hour, 12 hour, and 24 hour after drug administration
  clearance
volume of distribution | at Day 0: prior to drug administration (blank), then samples (5ml each) will be obtained at 0.5 hour, 1 hour, 1.5 hour, 2 hour, 2.5 hour, 3 hour, 4 hour, 5 hour, 6 hour, 8 hour, 10 hour, 12 hour, and 24 hour after drug administration
  volume of distribution
Detection of UGT2B7 SNPs (rs 7438135, rs 11740316) (genetic variation in Egyptian population) | 6 months
  Samples will be collected from each subject into tubes and stored at -80°C, Genomics DNA will be isolated according to manufactures instructions. Polymorphisms will be assessed using suitable recommended assay.

SECONDARY OUTCOMES:
Vital sign measurement following single dose administration as a measure of safety and tolerability | every month up to 6 months
  Vital sign measurements will include systolic and diastolic blood pressure
pulse rate | up to 6 months
  pulse rate
body temperature | up to 6-7 months
  body temperature measurement

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa A. Sabri, professor, Study Chair — Department of Clinical Pharmacy, Faculty of Pharmacy, Assiut University

REFERENCES:
- [Background] Reilly RF, Peixoto AJ, Desir GV. The evidence-based use of thiazide diuretics in hypertension and nephrolithiasis. Clin J Am Soc Nephrol. 2010 Oct;5(10):1893-903. doi: 10.2215/CJN.04670510. Epub 2010 Aug 26. PMID 20798254
- [Background] Psaty BM, Smith NL, Siscovick DS, Koepsell TD, Weiss NS, Heckbert SR, Lemaitre RN, Wagner EH, Furberg CD. Health outcomes associated with antihypertensive therapies used as first-line agents. A systematic review and meta-analysis. JAMA. 1997 Mar 5;277(9):739-45. PMID 9042847
- [Background] Campbell DB, Phillips EM. Short term effects and urinary excretion of the new diuretic, indapamide, in normal subjects. Eur J Clin Pharmacol. 1974 Oct 4;7(6):407-14. doi: 10.1007/BF00560352. No abstract available. PMID 4612998
- [Background] Wang TH, Hsiong CH, Ho HT, Shih TY, Yen SJ, Wang HH, Wu JY, Kuo BP, Chen YT, Ho ST, Hu OY. Genetic polymorphisms of metabolic enzymes and the pharmacokinetics of indapamide in Taiwanese subjects. AAPS J. 2014 Mar;16(2):206-13. doi: 10.1208/s12248-013-9535-x. Epub 2013 Dec 20. PMID 24357089